CLINICAL TRIAL: NCT01968486
Title: Reduced-fluence Verteporfin Photodynamic Therapy Plus Ranibizumab for Choroidal Neovascularization in Pathologic Myopia: 48 Weeks Study Results
Brief Title: Reduced-fluence Verteporfin Photodynamic Therapy Plus Ranibizumab for Choroidal Neovascularization in Pathologic Myopia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Chiosi Flavia, MD, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fidelio
Record Dates: First submitted 2013-07-10; First posted 2013-10-24 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Myopia, Degenerative
MeSH Terms: conditions — Myopia, Degenerative | interventions — Ranibizumab; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PDT Standard Fluence, ranibizumab (Experimental): verteporfin (6 mg/m2) SF (wavelength, 689 nm; dose, 50 J/cm2; light intensity, 600 milliwatt(mW)/cm2 for 83 s) plus 0.5 mg intravitreal ranibizumab
  Interventions: Drug: PDT standard fluence, ranibizumab
- PDT Reduced Fluence, ranibizumab (Experimental): verteporfin (6 mg/m2) RF ( wavelength, 689 nm; dose, 25 J/cm2 ; light intensity, 300 mW/cm2 for 83 s) plus 0.5 mg intravitreal ranibizumab
  Interventions: Drug: PDT reduced fluence, ranibizumab
- ranibizumab (Experimental): 0.5 mg (10 mg/ml) intravitreal ranibizumab.
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: PDT standard fluence, ranibizumab — In the verteporfin PDT combination therapy arm patients were treated on day one with 0.5 mg (10 mg/ml) IVR injection and after seven days with PDT standard fluence (wavelength, 689 nm; dose, 50 J/cm2; light intensity, 600 mW/cm2 for 83 s). Ranibizumab pro re nata (PRN) could be administered with a 30-day interval if re-treatment criterion were met. Re-treatment was based on increase of intraretinal or subretinal fluid > 50 μm on OCT; loss of 5 letters or more on BCVA Early Treatment Diabetic Retinopathy Study (ETDRS) chart; fluorescein leakage from the CNV on FA images.
  Other Names: Photodynamic therapy
  Arms: PDT Standard Fluence, ranibizumab
Drug: PDT reduced fluence, ranibizumab — In the verteporfin PDT combination therapy arm patients were treated on day one with 0.5 mg (10 mg/ml) IVR injection and after seven days with PDT reduced fluence ( wavelength, 689 nm; dose, 25 J/cm2 ; light intensity, 300 mW/cm2 for 83 s).Ranibizumab pro re nata (PRN) could be administered with a 30-day interval if re-treatment criterion were met. Re-treatment was based on increase of intraretinal or subretinal fluid > 50 μm on OCT; loss of 5 letters or more on BCVA Early Treatment Diabetic Retinopathy Study (ETDRS) chart; fluorescein leakage from the CNV on FA images.
  Other Names: Photodynamic therapy
  Arms: PDT Reduced Fluence, ranibizumab
Drug: ranibizumab — In the ranibizumab monotherapy arm patients were treated with a loading phase of three consecutive 0.5 mg (10 mg/ml) IVR injections every six weeks. Ranibizumab pro re nata (PRN) could be administered with a 30-day interval if re-treatment criterion were met. Re-treatment was based on increase of intraretinal or subretinal fluid > 50 μm on OCT; loss of 5 letters or more on BCVA Early Treatment Diabetic Retinopathy Study (ETDRS) chart; fluorescein leakage from the CNV on FA images.
  Other Names: Lucentis
  Arms: ranibizumab

SUMMARY:
To demonstrate the efficacy of ranibizumab in combination with reduced-fluence verteporfin photodynamic therapy (RF-PDT) in patients with subfoveal choroidal neovascularization secondary to pathologic myopia (PM).

DETAILED DESCRIPTION:
Sixty patients received ranibizumab 0.5 mg combined with reduced fluence (RF) verteporfin PDT. Ranibizumab was first administered to patients followed after seven days by RF-PDT. Subsequently intravitreal ranibizumab (IVR) was injected as needed (pro re nata). All patients were evaluated every 4 weeks for 48 weeks.

Main Outcome Measures: Mean change in best-corrected visual acuity (BCVA) from baseline at 48 weeks, reduced mean central foveal thickness (CFT) analyzed by optical coherence tomography (OCT) and improved macular sensitivity registered at microperimetry (MP) evaluation.

ELIGIBILITY:
Inclusion Criteria:

* pathologic myopia, defined as spherical equivalent greater than 6 D and axial length more than 26 mm (Carl Zeiss IOLMaster V 4.07; Carl Zeiss Meditec, Dublin, California, USA);
* posterior pole myopic retinal changes (posterior staphyloma, chorioretinal atrophy, papillary crescent);
* fluorescein angiography (FA) detection of the subfoveal or juxtafoveal CNV (CNV was classified as juxta-foveal if the lesion was closer than 200 mm but not under the geometric center of the foveal avascular zone);
* clear ocular media;
* duration of symptoms no longer than 4 weeks before enrollment.

Exclusion Criteria:

* prior treatment for CNV including previous intravitreal drugs injection or PDT-V;
* presence of other maculopathy as diabetic retinopathy or retinal vascular occlusion;
* history of recent myocardial infarction or other thromboembolic events;
* ongoing uncontrolled hypertension or glaucoma;
* refractive media opacities;
* eye surgery.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Mean change in best-corrected visual acuity (BCVA) from baseline | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Chiosi, MD, Principal Investigator — University of Campania Luigi Vanvitelli